CLINICAL TRIAL: NCT00096330
Title: Phase I Clinical Study of Folate
Brief Title: Folate-Depleted Diet Compared With Folate-Supplemented Diet in Preventing Colorectal Cancer in Patients at High Risk for Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000393455; P30CA016056 (NIH); RUH-PHO-0514-0404; RPCI-EPR-20703; AECM-0401022E; NEMCH-6060
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Diet Therapy; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: dietary intervention — oral folic acid supplementation once daily on days 57-84
Dietary Supplement: folic acid — oral folic acid supplementation once daily on days 1-56.

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain agents to try to prevent the development of cancer. The use of folic acid may be effective in preventing colorectal cancer. Eating a diet rich in folic acid may prevent the development of colorectal cancer.

PURPOSE: This randomized phase I trial is studying how well a folate-depleted diet works compared to a folate-supplemented diet in preventing colorectal cancer in patients who are at high risk for developing colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Analyze the effects of a folate-depleted vs a folate-supplemented diet on folate-related DNA endpoints (e.g., genomic and gene-specific DNA methylation and DNA strand breaks) in rectal epithelial cells in patients at high risk for colorectal neoplasia.
* Analyze the effects of these dietary interventions on folate-related DNA endpoints (e.g., genomic and gene-specific DNA methylation, DNA strand breaks, and uracil incorporation into DNA) in blood mononuclear cells in these patients.

Secondary

* Analyze the effects of these dietary interventions on the patterns of differential gene expression in rectal epithelial cells and blood mononuclear cells in these patients.

OUTLINE: This is a randomized, single-blind study.

* Run-in period: Patients are placed on an average folate-containing diet for 56 days.
* Randomization: After completion of the run-in period, patients are randomized to 1 of 2 arms.

  * Arm I (folate depleted diet): Patients are placed on a low-folate diet for 84 days. Patients receive oral folic acid supplementation once daily on days 57-84.
  * Arm II (folate supplemented diet): Patients continue on an average folate-containing diet for an additional 56 days. Patients receive oral folic acid supplementation once daily on days 1-56.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 20 patients (10 per arm) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy persons at increased risk for colorectal neoplasia due to 1 of the following reasons:

  * Personal history of colorectal adenomatous polyps
  * Family history of colorectal adenoma or adenocarcinoma
* No history of multiple family members with colorectal neoplasia that is suggestive of dominant hereditary neoplasia

PATIENT CHARACTERISTICS:

Age

* 40 to 72

Performance status

* Ambulatory

Life expectancy

* At least 6 months

Hematopoietic

* No excessive bleeding or coagulation disorder

Hepatic

* ALT or AST ≤ 2 times upper limit of normal
* No unexplained elevated alkaline phosphatase

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* Homocysteine concentration ≤ 17um/L
* No sustained blood pressure > 150/95 mm Hg for 3 consecutive readings

Other

* Vitamin B_12 ≥ 250 pg/mL
* Folate level ≤ 20 mg/dL
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No intestinal malabsorption or inflammatory bowel disease
* No prior malignancy except nonmelanoma skin cancer
* No calcium metabolism abnormalities or predisposing conditions, such as hyperparathyroidism
* No untreated hyperthyroidism
* No untreated insulin-requiring diabetes mellitus
* No daily alcohol intake > 2 ½ shot glasses of whiskey or three 8 ounce glasses of beer or wine
* No other serious illness that might limit life expectancy to < 6 months

PRIOR CONCURRENT THERAPY:

Biologic therapy

* None

Chemotherapy

* None

Endocrine therapy

* No concurrent hormone replacement therapy, including oral, transplanted, or injected contraceptives
* Concurrent thyroid hormone replacement is allowed as long as the patient is euthyroid for 3 months

Radiotherapy

* None

Surgery

* No prior gastrointestinal surgery, including gastrectomy or small or large bowel resections

  * Prior appendectomy or surgery of the esophagus allowed

Other

* More than 3 months since regular ingestion of ≥ 650 mg per day of aspirin (≥ 2 tablets of 325 mg regular strength OR > 1 tablet of 500 mg extra strength aspirin)
* More than 3 months since regular daily ingestion of nonsteroidal anti-inflammatory drugs
* At least 1 month since vitamin, mineral, or herbal supplementation
* No other concurrent vitamin, mineral, or herbal supplementation
* No concurrent anticoagulants
* No concurrent sterol-binding resins (i.e., cholestyramine)
* No other concurrent investigational drugs or medications that might alter rectal mucosal proliferation, folate metabolism, or renal/hepatic impairment
* No concurrent weight control medications
* No concurrent supplemental folate preparations containing > 400 mcg of folic acid per day
* No concurrent lipid-lowering medications

  * The following concurrent statin drugs are allowed provided patient has been taking a stable dose for ≥ 1 month:

    * Atorvastatin 10 or 20 mg/day
    * Fluvastatin 20 or 40 mg/day
    * Lovastatin 10 or 20 mg/day
    * Pravastatin 10 or 20 mg/day
    * Simvastatin 5 or 10 mg/day

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-09; Primary Completion 2007-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
•Analyze the effects of a folate-depleted vs a folate-supplemented diet on folate-related DNA endpoints | pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: James Marshall, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States